CLINICAL TRIAL: NCT06985368
Title: A Phase I Clinical Trial Evaluating the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of SIBP-A18 Injection in the Treatment of Advanced Malignant Solid Tumor Patients
Brief Title: A Clinical Trial of SIBP-A18 Injection in the Treatment of Advanced Malignant Solid Tumor Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIBP-A18-I
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor Malignancy
Keywords: Solid Tumor Malignancy; ADC; Safety; Efficacy; Pharmacokinetics

STUDY DESIGN:
Intervention Model Description: This study is an open, multi dose increasing single and multiple dose study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIBP-A18 (Experimental): The participants enrolled will be sequentially assigned to the corresponding dose level.
  Interventions: Drug: SIBP-A18

INTERVENTIONS:
Drug: SIBP-A18 — SIBP-A18 formulation for injection, Claudin18.2-ADC. Strength: 1.0, 2.0, 3.2, 4.0, 4.8, 5.6, 6.4 and 8.0 mg/kg. Intravenous infusion administration, with a treatment cycle of every 21 days, administered once on the first day of each cycle. The dose escalation stage, 1mg/kg and 2mg/ kg were subjected to accelerated titration, where the safety was evaluated within 21 days after the first administration to one participant. If dose-limiting toxicity (DLT) occurred, the traditional "3+3" dose escalation method was immediately switched. If DLT does not occur, the next dose group will be explored. The third stage will use RP2D for further exploration.

SUMMARY:
The main purpose To evaluate the safety, tolerability, and pharmacokinetic characteristics of SIBP-A18 and determine the maximum tolerable dose (MTD) and phase II recommended dose (RP2D).

A secondary purpose To preliminarily evaluate the anti-tumor efficacy of SIBP-A18. Evaluate the effect of SIBP-A18 injection on Q to T interval/Corrected QT interval (QT/QTc interval) in participants with advanced solid tumors

DETAILED DESCRIPTION:
This study is an open, multi-dose increasing single and multiple doses increasing, dose expanding, and indication expanding study to evaluate the safety, tolerability, pharmacokinetics, immunogenicity, preliminary anti-tumor efficacy, and explore potential biomarkers of SIBP-A18 in patients with advanced solid tumors.

This study is divided into three stages and is planned to be set up eight dose groups, including 1.0, 2.0, 3.2, 4.0, 4.8, 5.6, 6.4 and 8.0 milligram per kilogram (mg/kg). The first stage is the dose escalation stage, which will start from the first and second doses for enrollment. If necessary, a 3+3 dose escalation design will be used. The second stage is the dose expansion stage, where two or more doses are selected to enter the dose expansion phase, and 6-9 participants will be enrolled in each dose group for dose expansion. The third stage is the indication expansion stage, where RP2D is preliminarily determined based on the escalation and expansion of dosage in the early stage. Using RP2D for indication expansion, we plan to expand three indication cohorts, with at least 30 participants selected for each cohort.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 18 to 75 years old (including boundary values), regardless of gender.
* The clinical diagnosis of enrolled participants should meet the following criteria:

  1. Dose escalation and dose expansion stage: Patients with advanced solid tumor diagnosed by histology and/or cytology, who have previously failed standard treatment, lack standard treatment regimens, are intolerant to standard treatment, or are currently not eligible for standard treatment.
  2. Indications expansion stage:

Queue 1: CLDN18.2 positive late stage gastric cancer/gastroesophageal junction cancer (GC/GEJC) confirmed by histology or cytology with standard treatment failure, intolerance, or no standard treatment.

Queue 2: Late stage CLDN18.2 positive PC confirmed histologically or cytologically with standard treatment failure, intolerance, or no standard treatment.

Queue 3: CLDN18.2 positive late biliary tract cancer (BTC) confirmed histologically or cytologically with standard treatment failure, intolerance, or no standard treatment.

* Willing and able to provide sufficient fresh collected or archived tumor tissue samples within two years.
* At least one measurable lesion must be selected as the target lesion (according to Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 standard, computed tomography (CT) or magnetic resonance imaging (MRI)) (for lesions that have previously received radiotherapy, only with clear progression can they be selected as the target lesion).
* The patient has not previously received any form of topoisomerase I inhibitor in the past, including antibody drug conjugates
* ECOG score 0-1.
* Expected survival time ≥ 3 months.
* During the screening period, the main organ functions were basically normal (no medical support such as blood transfusion, granulocyte colony-stimulating factor (G-CSF), or other medical support was received within 14 days before the use of the investigational drug):

Blood routine: Absolute value of neutrophils (NE #) ≥ 1.5 × 10^9/L, platelet (PLT) count

≥ 90 × 10 9/L, hemoglobin (HGB) ≥ 90 g/L.

* Women of childbearing age during the screening period who have a negative blood pregnancy test and are capable of reproduction (including male participants) have no pregnancy plan and voluntarily take effective contraceptive measures during the trial period and within 6 months after the last dose.
* Voluntarily participate in this study and sign an informed consent form.

Exclusion Criteria:

* Participants with the following tumors:

  * The participant has had other malignant tumors that have not been cured within the past 5 years (excluding malignant tumors that have been clearly cured, such as thyroid cancer, cured basal cell carcinoma of the skin, and cervical carcinoma in situ).
  * The participant has untreated imaging confirmed central nervous system metastasis.
  * Meningeal metastases.
  * Patients with brain metastases who have received systematic or curative brain metastasis treatment (radiotherapy or surgery) in the past, have been confirmed stable by imaging for at least 4 weeks, and have stopped systemic hormone, antiepileptic, convulsive drugs, and other treatments for more than 2 weeks without clinical symptoms can be enrolled.
* Participants with a history of previous treatment or surgery, or those who received the following anti-tumor treatments during the planned trial period:

  * Patients who accepted the instructions clearly containing traditional Chinese patent medicines and simple preparations with anti-tumor effect within 2 weeks before the first administration;
  * Patients undergoing adjuvant therapy within 6 months after surgery;
  * Patients who have not recovered from the toxicity of the previous anti-tumor treatment to normal or ≤ level 1 (excluding hair loss);
  * Patients who have undergone major surgery, radiation therapy, biological therapy, or chemotherapy within 4 weeks prior to their first administration, or who have received systemic treatment such as unhealed surgical wounds, ulcers or fractures, or other clinical trial drugs.
  * Patients who plan to receive any other anti-tumor treatment (chemotherapy, radiation therapy, immunotherapy, cytokine therapy other than erythropoietin) during the trial period should be excluded (excluding testosterone lowering therapy for prostate cancer patients).
  * The dose (prednisone>10 mg/d or equivalent) at which immunosuppressive effects are achieved by receiving immunosuppressive agents or systemic corticosteroids within one week prior to the use of the investigational drug.
* Participants with a history of previous illnesses or laboratory tests that show the following abnormalities:

Individuals with abnormal coagulation function and a tendency to bleed, or who are undergoing thrombolysis or anticoagulation treatment or have lost blood or donated more than 400 mL within 2 months prior to administration.

* Have a history of immunodeficiency, including HIV testing positive, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation.
* Have a clear history of neurological or psychiatric disorders, including epilepsy or dementia.

  * Screening period for syphilis spiral antibody positive individuals; Individuals with active hepatitis B virus (HBV) and hepatitis C virus (HCV) infections; Except those with stable hepatitis B (DNA titer below the lower detection limit) and cured hepatitis C (HCV RNA test negative) after drug treatment.
  * Patients with ascites, pleural effusion, and pericardial effusion accompanied by clinical symptoms during the screening period who require drainage, or those who have undergone serous cavity drainage within 4 weeks before the first administration.
  * The screening period is accompanied by severe, progressive, or uncontrollable diseases, and the researcher's evaluation determines that the participation of the participants in the study will increase the risk. Including but not limited to:
* Cerebrovascular accidents or transient ischemic attacks (within the first 6 months of screening); Suffering from heart disease judged by the researcher as unsuitable for participation in this trial, with a severity of cardiac or renal dysfunction ≥ Level II.

  * According to the researcher's judgment, there are accompanying diseases that seriously endanger patient safety or affect patient completion of the study.

    1. Hypertension that cannot be controlled clinically.
    2. Diabetes with poor drug control.
    3. Clinically significant thyroid diseases judged by researchers as unsuitable for inclusion.
    4. Serious infections that occurred within 4 weeks prior to initiating research treatment.
  * Individuals with a history of severe allergies to protein products, Chinese hamster ovary cell (CHO) cell products, and other recombinant human or humanized antibodies, or to the components of the investigational drug.
  * Pregnant and lactating women.
  * Patients deemed unsuitable for inclusion by researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2028-05-15 (Estimated); Study Completion 2028-09-15 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) | From day 1 after the first dose to day 28 after the last dose
  That is adverse events, any adverse events that occurred to the participant during the study period.
Serious Adverse Events (SAE) | From day 1 after the first dose to day 28 after the last dose
  That is serious adverse events, any serious adverse events that occurred to the participant during the study period.
Area Under The Plasma Concentration Versus Time Curve (AUC) | Day 1, Day 22 and Day 63 after the first dose
  It shows the degree to which a drug is absorbed and used in the body.
Peak Plasma Concentration (Cmax) | Day 1, Day 22 and Day 63 after the first dose
  It shows the highest plasma concentration of a drug that can be achieved after administration.
Peak Time (Tmax) | Day 1, Day 22 and Day 63 after the first dose
  That is peak time of drug action, it shows the time required to reach the maximum concentration on the participant plasma concentration curve after administration.
Terminal elimination half-life (T ½ ) | Day 1, Day 22 and Day 63 after the first dose
  It reflects how quickly the drug is eliminated from the body.
Clearance Rate (CL) | Day 1, Day 22 and Day 63 after the first dose
  Apparent volume of drug distribution removed from the body per unit time.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 6 weeks after the last evaluation
  The proportion of participants whose tumor volume shrinks to a predetermined value and maintains the minimum time limit and is the sum of complete and partial responses.
Disease control rate (DCR) | 6 weeks after the last evaluation
  In clinical trials, the percentage of participants with advanced cancer who responded fully to cancer treatment, partially responded, and had stable disease.
Progression-free survival (PFS) | 6 weeks after the last evaluation
  The time between the onset of randomization and the onset (of any aspect) of tumor progression or death (from any cause).
overall survival (OS) | 6 weeks after the last evaluation
  From randomization to time of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Huang, Docter, Principal Investigator — Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No